CLINICAL TRIAL: NCT06628934
Title: Wearable Sensors for Quantitation of Impaired Gait and Balance
Brief Title: Wearable Gait Sensors
Status: Active, not recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB17-0253
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Spinocerebellar Ataxia
MeSH Terms: conditions — Spinocerebellar Ataxias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spinocerebellar Ataxia: Individuals with genetically-confirmed diagnosis of SCA
- Healthy Controls: Healthy Controls

SUMMARY:
This research study is testing body-worn sensors to measure movement during simple tests of coordination, in order to evaluate the progression and severity of Spinocerebellar ataxia.

DETAILED DESCRIPTION:
Study participants will complete a neurological exam with sensors (iSARA exam) and three patient-reported questionnaires (PROM-Ataxia, ABC Scale, EQ-5D-5L). Participation will take about an hour.

ELIGIBILITY:
Inclusion Criteria:

* Ataxia Group - Individuals who have a genetic-confirmation of SCA diagnosis and are able to sit or stand unassisted for 30 seconds and follow directions.
* Healthy Control Group - Individuals who are able to sit or stand unassisted for 30 seconds and follow directions.

Exclusion Criteria:

* Any other neurological or musculoskeletal disorder not attributed to the SCA that could affect balance, gait or voluntary movement.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of Ataxia Clinics
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-06-23 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
iSARA | 8 Years
  Digital measurements collected by wearable inertial sensors during instrumented Scale for the Assessment and Rating of Ataxia (iSARA).

SECONDARY OUTCOMES:
Patient Reported Outcome Measure of Ataxia (PROM-Ataxia) | 8 Years
  Comparing patient-reported outcome measures evaluation of severity and progression to the measurements collected by wearable inertial sensors during instrumented Scale for the Assessment and Rating of Ataxia (iSARA). The PROM-Ataxia is a 70-item assessment of physical, mental health, and activities of daily living, each scored on a 0-4 Likert scale. Scores are totaled.
Activities-specific Balance Confidence (ABC) Scale | 8 Years
  Comparing patient-reported outcome measures evaluation of severity and progression to the measurements collected by wearable inertial sensors during instrumented Scale for the Assessment and Rating of Ataxia (iSARA). The ABC scale is a 16 item scale with a rating scale from 0 (no confidence) to 100 (complete confidence) in avoiding a fall. The score is determined by taking the average of all items.
EQ-5D-5L | 8 Years
  Comparing patient-reported outcome measures evaluation of severity and progression to the measurements collected by wearable inertial sensors during instrumented Scale for the Assessment and Rating of Ataxia (iSARA). The EQ-5D-5L is a 5 item descriptive system to describe current mobility, self-case, usual activities, pain/discomfort, and anxiety/depression.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No